CLINICAL TRIAL: NCT02715388
Title: Proof of Concept - Digital Electro-optical Surgical Platform as Replacement for Operational Microscopes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elbit Systems LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0389-15-TLV
Record Dates: First submitted 2016-03-15; First posted 2016-03-22 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Retinal Detachment
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silicon oil removal 3D visualization (Experimental)
  Interventions: Device: GlasScope Surgical Microscope

INTERVENTIONS:
Device: GlasScope Surgical Microscope — 3D visualization of the poterior chamber for silicon oil removal

SUMMARY:
Evaluate the use of Elbit's digital electro-optical systems for generating detailed high quality video imaging during surgery, and thus improving the surgeon's visualization, performance and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18.
* Pseudophakia patients with silicone oil in the vitreous cavity.
* Silicone oil density of 1500 centistoke or 5500 CS.
* Good corrected visual acuity (> 6/10) in the second eye.
* Lack of additional ocular pathology that would reduce the quality of vision during surgery (corneal scar, Posterior Capsular Opacity, low transmission in the implantable lens, non-expanded pupil).

Exclusion Criteria:

* Additional ocular pathology that would reduce the quality of vision during surgery (corneal scar, Posterior Capsular Opacity, low transmission in the implantable lens, non-expanded pupil).
* The presence of heavy silicone oil (OXANE) in the vitreous cavity.
* Posterior segment pathology in the second eye.
* Special populations (children under the age of 18, pregnant women)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01; Primary Completion 2022-01 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Field of view of GlasScope surgical microscope | Up to 3 days after surgery
Depth of field of GlasScope surgical microscope | Up to 3 days after surgery
3D perception of GlasScope surgical microscope | Up to 3 days after surgery
  3D perception of GlasScope surgical microscope is assessed by the surgeon ability to perform surgical gentle procedures using the surgical tools on the eye tissues - both inner and posterior parts of the eye.

SECONDARY OUTCOMES:
Surgeon fatigue and neck strain (questionnaire) | Up to 7 days after surgery
  Questioning the surgeons after surgery on the pain and stress during the use of Glasscope causing decreased performance/lack of concentration/fatigue, the complexity on keeping the eye-piece image in the surgeon sight, how the instrument prevents the surgeon situation awareness in the operating room, the stress and fatigue on the surgeon eyes for long duration of observation in the image

CONTACTS AND LOCATIONS:
Overall Officials: Adiel Barak, Prof, Principal Investigator — Head of Retina Department, Sourasky Medical Center
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No